CLINICAL TRIAL: NCT00724945
Title: Comparison of Two Soft Bifocal Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CR-1485CK
Record Dates: First submitted 2008-07-25; First posted 2008-07-30 (Estimated); Results first posted 2010-01-27 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Presbyopia
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- senofilcon A / balafilcon A (Active Comparator): senofilcon A multifocal lenses worn first, balafilcon A multifocal lenses worn second
  Interventions: Device: balafilcon A; Device: senofilcon A
- balafilcon A/senofilcon A (Active Comparator): balafilcon A multifocal lenses worn first, senofilcon A multifocal lenses worn second
  Interventions: Device: balafilcon A; Device: senofilcon A

INTERVENTIONS:
Device: balafilcon A — multifocal contact lens
Device: senofilcon A — multifocal contact lens

SUMMARY:
The purpose of the study is to compare the visual performance of two soft bifocal contact lenses.

ELIGIBILITY:
Inclusion Criteria:

* The subject must between 35 and 70 years of age.
* The subject must have presbyopic symptoms or be already wearing presbyopic contact lens correction.
* The subject's spherical equivalent distance refraction must be in the range of -1.00 to -6.00 or -9.00 to -10.00 in each eye.
* Refractive cylinder must be -0.75 D in each eye.
* The subject must have an ADD power of +0.75D to +2.50D in each eye.
* The subject must have best corrected visual acuity of 20/20-3 or better in each eye
* The subject's must have at least 20/30-distance vision OU with the study contact lenses.
* The subject must agree that they are comfortable with their vision prior to being dispensed the study lenses
* The subject must be an adapted soft contact lens wearer in both eyes.
* The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol.
* The subject must read and sign the STATEMENT OF INFORMED CONSENT and be provided a copy of the form.

Exclusion Criteria:

* Ocular or systemic allergies or disease that may interfere with contact lens wear.
* Systemic disease, autoimmune disease or use of medication, which may interfere with contact lens wear.
* Clinically significant (grade 3 or 4) corneal edema, corneal vascularization, corneal staining or any other abnormality of the cornea, which may contraindicate contact lens wear
* Clinically significant (grade 3 or 4) tarsal abnormalities that might interfere with contact lens wear.
* Any ocular infection.
* Any corneal distortion resulting from previous hard or rigid gas permeable contact lens wear.
* Pregnancy or lactation
* Any infectious disease (e.g., hepatitis, tuberculosis) or an immunosuppressive disease (e.g., HIV).
* History of diabetes
* History of binocular vision abnormality or strabismus

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2008-07; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Dr. James Weber & Associates, Jacksonville, Florida
  - Ted Brink & Associates, Jacksonville, Florida
  - Jacksonville, Florida
  - Eye Associates of Winter Park, Winter Park, Florida
  - Lee Rigel, East Lansing, Michigan
  - Timothy R. Poling, OD, Roanoke, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Senofilcon A/Balafilcon A: senofilcon A multifocal contact lenses worn first, balafilcon A multifocal contact lenses worn second
- Balafilcon A/Senofilcon A: balafilcon A multifocal contact lenses worn first/ senofilcon A multifocal contact lenses worn second
Period: Period 1
Arm/Group | Senofilcon A/Balafilcon A | Balafilcon A/Senofilcon A
Started | 58 | 55
Completed | 55 | 54
Not Completed | 3 | 1
Not completed — non-compliance | 1 | 0
Not completed — Adverse Event | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Period: Period 2
Arm/Group | Senofilcon A/Balafilcon A | Balafilcon A/Senofilcon A
Started | 55 | 54
Completed | 51 | 54
Not Completed | 4 | 0
Not completed — lens comfort issue | 3 | 0
Not completed — lens physiology issue | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall: The reporting group for baseline characteristics includes all subjects that completed the study wearing contact lenses made from either senofilcon A or balafilcon A material. Excluded are 8 subjects that discontinued and 2 subjects dispensed lenses from outside study contact lens materials.
Arm/Group | Overall
Number analyzed (Participants) | 103
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.2 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87
  Male | 16
Region of Enrollment [Number; unit: participants]
  United States | 103

OUTCOME MEASURES:

1. Primary Outcome: Distance Visual Acuity
Description: This outcome measures vision while subjects are looking at objects in the distance and is measures in logMARs.logMAR is the logarithm of the minimum angle of resolution.The ideal is 0.0 and represents 20/20 Snellen acuity.logMAR values >0.00 indicate vision poorer than ideal and values<0.0 indicate vision greater than ideal
Time Frame: after 1 week of wear
Population: Analysis includes participants who completed the study per protocol.
Measure: Least Squares Mean (Standard Error); unit: logMAR units
Arm/Group | Senofilcon A | Balafilcon A
Number analyzed (Participants) | 103 | 103
logMAR units | -0.08591 (0.008816) | -0.10267 (0.008855)
Statistical Analysis 1: Comparison: Senofilcon A; Alternative hypothesis: senofilcon A multifocal would be better than or equal to 0.1 logMAR units; Test type: Superiority or Other; Mixed Models Analysis; Least Square Mean = -0.08591, 95% CI [-0.08591 to -0.06857], Standard Error of Mean 0.008816

2. Primary Outcome: Near Visual Acuity
Description: This outcome measures vision while subjects are looking at objects near to them and is measured in logMARs. logMAR is the logarithm of the minimum angle of resolution.The ideal is 0.0 and represents 20/20 Snellen acuity.logMAR values >0.00 indicate vision poorer than ideal and values<0.0 indicate vision greater than ideal.
Time Frame: after 1 week wear
Measure: Least Squares Mean (Standard Error); unit: logMAR units
Arm/Group | Senofilcon A | Balafilcon A
Number analyzed (Participants) | 103 | 103
logMAR units | 0.02711 (0.008816) | 0.01933 (0.008861)
Statistical Analysis 1: Comparison: Senofilcon A; Alternative hypothesis: senofilcon A multifocal lens would be better than or equal to 0.17 logMAR units; Test type: Superiority or Other; Mixed Models Analysis; Least Square Mean = 0.02711, 97.5% CI [0.02711 to 0.04445], Standard Error of Mean 0.008816

3. Primary Outcome: Subject Vision
Description: Subjects responded to "How would you rate the overall quality of vision with these study contact lenses" using the following scale: 1=poor, 2=fair, 3=good, 4=very good, 5=excellent.
Time Frame: after 1 week wear
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Senofilcon A | Balafilcon A
Number analyzed (Participants) | 103 | 103
Scores on a scale | 3.4594 (0.09926) | 3.3853 (0.09926)
Statistical Analysis 1: Comparison: Senofilcon A vs Balafilcon A; Alternative hypothesis: senofilcon A multifocal lens will have subjective vision that is non-inferior to balafilcon A multifocal; Test type: Non-Inferiority or Equivalence — The non-inferiority margin is -0.5; Mixed Models Analysis; Mean Difference (Final Values) = 0.07407, 97.5% CI [-0.1797 to 0.07407], Standard Error of Mean 0.1279 — Mean difference was calculated as senofilcon A multifocal minus balafilcon A multifocal

ADVERSE EVENTS:
Arm/Group | Senofilcon A/Balafilcon A | Balafilcon A/Senofilcon A
Serious Adverse Events (participants affected / at risk) | 0/58 | 0/55
Other Adverse Events (participants affected / at risk) | 0/58 | 0/55

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI may not publish, divulge, reveal, disclose, or use the data and or results of the study without prior written consent of Vistakon.